CLINICAL TRIAL: NCT01967186
Title: Open Multi-Center Randomized Study to Compare Safety and Efficacy of Islet Transplantation Using The Intraportal or Intramuscular Site in Simultaneous Islet and Kidney Transplantation
Brief Title: Intraportal or Intramuscular Site for Islets in Simultaneous Islet and Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Nordic Network For Clinical Islet Transplantation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIK01
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Type 1 Diabetes; End Stage Renal Disease
Keywords: Type 1 diabetes; islets; transplantation; nephropathy; intramuscular
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Failure, Chronic; Kidney Diseases | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intraportal islet transplantation (Experimental): Subject randomized to the protocol with intraportal islet transplantation and kidney transplantation
  Interventions: Procedure: Intraportal islet transplantation; Procedure: Kidney transplantation
- Intramuscular islet transplantation (Experimental): Subject randomized to the protocol with intramuscular islet transplantation and kidney transplantation
  Interventions: Procedure: Intramuscular islet transplantation; Procedure: Kidney transplantation
- Intramuscular transpl with stemcells (Experimental): Subject randomized to the protocol with intramuscular islet transplantation and where islets have been incubated autologous mesenchymal stemcells. Will also receive kidney transplant
  Interventions: Procedure: Intramuscular transpl with stemcells; Procedure: Kidney transplantation
- Kidney transplantation only (Active Comparator): Subject that only undergoes kidney transplantation
  Interventions: Procedure: Kidney transplantation

INTERVENTIONS:
Procedure: Intraportal islet transplantation
  Arms: Intraportal islet transplantation
Procedure: Intramuscular islet transplantation
  Arms: Intramuscular islet transplantation
Procedure: Intramuscular transpl with stemcells
  Arms: Intramuscular transpl with stemcells
Procedure: Kidney transplantation — All patients will undergo kidney transplantation regardless of arm

SUMMARY:
Islet transplantation is a promising treatment of type 1 diabetes in selected cases. Results are however hampered by a relatively low number of islets surviving the transplantation into the liver, which currently is the site for transplantation. In the present study we compare a new transplantation site (intramuscular in the arm) to the golden standard (the liver) in patients undergoing kidney transplantation from the same donor. In half of the intramuscular transplanted patients, the islets will be mixed with mesenchymal stemcells from the recipient to, possibly, improve the immunological aspects of the transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 65 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years at the time of enrolment.
* Absence of stimulated C-peptide <0.1 nmol/L in response to a MMTT.
* All subjects must have received adequate medical treatment of their diabetes under the guidance from an experienced diabetologist.
* All subjects must have renal failure and be eligible for renal transplantation according to local criteria.

Exclusion Criteria:

* Patients with prior organ transplants
* Patients that qualify for local simultaneous pancreas-kidney transplantation program and who prefer that option
* Patients with body mass index BMI > 28.
* Insulin requirement > 1 Unit/kg/day. If the patient is on peritoneal dialysis the same limit is set when the extra carbohydrates in the dialysis fluids have been accounted for.
* Consistently abnormal liver function tests ( > 1.5 x the upper limit of normal on two consecutive measurements > 2 weeks apart)
* Unstable diabetic retinopathy
* Hypercoagulability disorder or coagulopathy or International normalized ratio (INR)>1.5
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Patients with unstable cardiovascular status
* Patients with active infections, unless treatment is not judged necessary by the investigators
* Patients with serological evidence of infection with HIV, hepatitis B (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
C-peptide derived from the Mixed Meal Tolerance Test (MMTT) | 365 days (+/-14) after kidney transplantation
  Percentage of patients in each study group reaching a systemic C-peptide derived from the MMTT above 0.1 nmol/L basal (fasting) and 90-min 0.3 nmol/L 75 (+/-5) and 365 days (+/-14) after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Kaija Salmela, MD PhD, Principal Investigator — Kidney Transplant Unit, Helsinki University Hospital, Helsinki, Finland